CLINICAL TRIAL: NCT00347958
Title: Safety Among Adolescents and Adults of Revaccination With Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (Adacel®) 4 to 5 Years After a Previous Dose
Brief Title: Descriptive, Open-label, Multicenter Study of the Safety of Redosing With ADACEL® Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TD518
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Results first posted 2010-07-22 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Tetanus; Diphtheria; Pertussis
Keywords: Tetanus,; Diphtheria,; Pertussis
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough | interventions — Vaccines; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adacel vaccine group (Experimental): Participants 15 to 69 years of age who received a dose of Adacel vaccine in one of three previous studies (Td501, or Td502, or Td505), revaccinated in Study Td518.
  Interventions: Biological: Tetanus-diphtheria-acellular pertussis (Tdap) vaccine

INTERVENTIONS:
Biological: Tetanus-diphtheria-acellular pertussis (Tdap) vaccine — 0.5mL, Intramuscular (IM)
  Other Names: Adacel®

SUMMARY:
Objectives:

To provide safety data on revaccination with ADACEL® vaccine.

To describe the immune response to tetanus, diphtheria, and pertussis antigens following revaccination with ADACEL® vaccine 4-5 years after first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Previously received ADACEL vaccine as part of Aventis Pasteur studies Td501, Td502, or Td505.
* At least 15 but no greater than 69 years of age at the time of vaccination in this trial.
* Signed Institutional Review Board (IRB)-approved informed assent / consent form.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman, inability to become pregnant or negative serum/urine pregnancy test.

Exclusion Criteria:

* Any condition which, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Serious chronic disease (ie, cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric) that is unstable or that might:

  * interfere with the ability to participate fully in the study; or
  * interfere with evaluation of the vaccine.
* Known or suspected impairment of immunologic function.
* Febrile illness within the last 72 hours or an oral temperature ≥100.4°F (≥38°C) at the time of inclusion.
* History of documented tetanus, diphtheria or pertussis disease within the preceding 5 years.
* Known or suspected receipt of a tetanus-, diphtheria- or pertussis-containing vaccine since participation in Study Td501, Td502, or Td505. (Receipt of Menactra vaccine at any time prior to the present study is permitted, subject to the next exclusion criterion).
* Received any vaccine, other than influenza vaccine, in the 28-day period prior to enrollment or scheduled to receive any vaccine, other than influenza vaccine, in the 28-day period after enrollment. For influenza vaccine only, defer if received in the 14-day period prior to enrollment or scheduled to receive in the 14-day period after enrollment
* Administration of immune globulin or other blood products within the last three months, or injected or oral corticosteroids or other immunomodulator therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting less than 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Suspected or known hypersensitivity to any of the vaccine components or to latex.
* Unable to attend the scheduled visits or to comply with the study procedures.
* In females of childbearing potential, a positive or equivocal urine pregnancy test at enrollment.
* Nursing mother.
* Participation in another interventional clinical trial in the 4 weeks preceding enrollment or planning to participate in another interventional clinical trial during the planned period of this study.
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial visits or procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular (IM) vaccination.
* Subject deprived of freedom by an administrative or court order, or under the stress of an emergency setting, or hospitalized without his/her consent.

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (10):
- United States (4):
  - Jonesboro, Arkansas
  - Bossier City, Louisiana
  - University Heights, Ohio
  - Pittsburgh, Pennsylvania
- Canada (6):
  - Coquitlam, British Columbia
  - Surrey, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Beauport, Quebec
  - Montreal, Quebec

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 21 August 2006, to 12 April 2007, in 6 clinical centers in the US and 6 clinical centers in Canada.
Pre-assignment Details: A total of 545 participants were enrolled and vaccinated in the study. Data on 544 participants that met the inclusion and exclusion criteria were analyzed and reported. One participant who did not receive Adacel® vaccine in one of the previous studies was excluded from the Safety Analysis Set.
Groups:
- Adacel® Vaccine Group: Participants 15 to 69 years of age who received a dose of Adacel vaccine in one of three previous studies (Td501, or Td502, or Td505), revaccinated in Study Td518.
Period: Overall Study
Arm/Group | Adacel® Vaccine Group
Started | 544
Completed | 540
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adacel® Vaccine Group
Number analyzed (Participants) | 544
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 169
  Between 18 and 65 years | 368
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284
  Male | 260
Region of Enrollment [Number; unit: participants]
  United States | 194
  Canada | 350

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Solicited Injection Site and Systemic Reactions Post-Vaccination
Description: Solicited Injection Site Reactions: Pain, Erythema/Redness, Swelling. Solicited Systemic Reactions: Fever (Temperature), Headache, Myalgia, Malaise.
Time Frame: 0-14 days post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
  The solicited systemic reaction, malaise was not collected in the previous studies.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adacel® Vaccine Group
Number analyzed (Participants) | 544
Percentage of Participants
  Any Solicited Injection Site Reaction | 89
  Any Injection Site Pain | 88
  Grade 3 Injection Site Pain (Incapacitating) | 2
  Any Injection Site Erythema/Redness | 29
  Grade 3 Injection Site Erythema/Redness (≥ 5 cm) | 3
  Any Injection Site Swelling | 26
  Grade 3 Injection Site Swelling (≥ 5 cm) | 3
  Any Fever | 7
  Grade 3 Fever (> 39.0 ºC or > 102.2 ºF) | 1
  Any Headache | 53
  Grade 3 Headache (Prevents daily activities) | 3
  Any Myalgia | 61
  Grade 3 Myalgia (Prevents daily activities) | 4
  Any Malaise | 38
  Grade 3 Malaise (Prevents daily activities) | 3

2. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Tetanus and Diphtheria Antibodies Pre- and Post-Vaccination.
Description: Pre- and post-vaccination GMTs and their 95% confidence intervals for diphtheria were determined by toxin neutralization testing; the other antibody levels were determined by enzyme-linked immunosorbent assay testing.
Time Frame: Day 28 post-vaccination
Population: Geometric mean titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adacel® Vaccine Group
Number analyzed (Participants) | 451
Titers
  Tetanus (IU/mL) Pre-Dose, n = 445 | 1.41 [1.27 to 1.56]
  Tetanus (IU/mL) Post-Dose, n = 445 | 9.62 [9.06 to 10.2]
  Diphtheria (IU/mL) no Menactra Pre-Dose, n = 379 | 0.133 [0.110 to 0.162]
  Diphtheria (IU/mL) no Menactra Post-Dose n = 379 | 2.17 [1.84 to 2.56]
  Diphtheria (IU/mL) with Menactra Pre-Dose n = 64 | 4.45 [2.77 to 7.15]
  Diphtheria (IU/mL) with Menactra Post-Dose n = 64 | 8.70 [6.59 to 11.5]

3. Other Pre Specified Outcome: Geometric Mean Titers (GMTs) of Pertussis Antibodies Pre- and Post-Vaccination.
Description: Pre- and post-vaccination GMTs and their 95% confidence intervals for Pertussis were determined by enzyme-linked immunosorbent assay testing.
Time Frame: Day 28 post-vaccination
Population: Geometric mean titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Adacel® Vaccine Group
Number analyzed (Participants) | 451
Titers
  Pertussis PT (EU/mL) Pre-Dose, n = 381 | 21.3 [19.4 to 23.5]
  Pertussis PT (EU/mL) Post-Dose, n = 425 | 104 [97.0 to 112]
  Pertussis FHA (EU/mL) Pre-Dose, n = 450 | 34.6 [31.9 to 37.5]
  Pertussis FHA (EU/mL) Post-Dose, n = 450 | 201 [189 to 215]
  Pertussis PRN (EU/mL) Pre-Dose, n = 451 | 37.3 [32.7 to 42.6]
  Pertussis PRN (EU/mL) Post-Dose, n = 451 | 218 [201 to 236]
  Pertussis FIM (EU/mL) Pre-Dose, n = 445 | 165 [145 to 187]
  Pertussis FIM (EU/mL) Post-Dose, n = 450 | 749 [697 to 806]

4. Other Pre Specified Outcome: Percentage of Participants With Tetanus and Diptheria Antibody Titers ≥ 0.1 Pre- and Post-Vaccination With Adacel®
Description: Seroprotection: Tetanus or diphtheria titer ≥ 0.1 after Adacel® vaccination. Tetanus titers determined by enzyme-linked immunosorbent assay; diphtheria titers determined by toxin neutralization assay.
Time Frame: Day 28 post-vaccination
Population: Tetanus and diphtheria antibody analyses were in all enrolled and vaccinated participants in the per-protocol population. Diphtheria antibody titers were analyzed separately for participants without and with an intervening Menactra vaccination between the previous study and Study Td518.
Measure: Number; unit: Percentage of Participants
Arm/Group | Adacel® Vaccine Group
Number analyzed (Participants) | 451
Percentage of Participants
  Tetanus (IU/mL) Pre-Dose | 96
  Tetanus (IU/mL) Post-Dose | 100
  Diphtheria (IU/mL) without Menactra, Pre-Dose | 61
  Diphtheria (IU/mL) without Menactra, Post-Dose | 95
  Diphtheria (IU/mL) Menactra, Pre-Dose | 95
  Diphtheria (IU/mL) Menactra, Post-Dose | 100

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to 6 months post-vaccination
Arm/Group | Adacel® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 7/544
Other Adverse Events (participants affected / at risk) | 479/544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adacel® Vaccine Group (N=544)
Cardiac arrest (Cardiac disorders) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0)
Pyelonephritis (Metabolism and nutrition disorders) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Carcinoid tumour of the appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Adacel® Vaccine Group (N=544)
Nasopharyngitis (Infections and infestations) | 44 (45)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 35 (40)
Injection site pain (General disorders) | 472/539 (472)
Injection site erythema/redness (General disorders) | 154/539 (154)
Injection site swelling (General disorders) | 138/539 (138)
Pyrexia (Fever) (General disorders) | 35/538 (35)
Headache (Nervous system disorders) | 287/539 (287)
Malaise (General disorders) | 206/539 (206)
Myalgia (Musculoskeletal and connective tissue disorders) | 329/539 (329)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications